CLINICAL TRIAL: NCT02340650
Title: High Resolution Imaging for Early and Better Detection of Bladder Cancer
Acronym: HRME_Bladder
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Principal Investigator, Nadeem N Dhanani, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0144
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Bladder Cancer
Keywords: suspicious bladder lesion, normal bladder tissue
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bladder Cancer Patients: High resolution images of normal bladder tissue and suspicious bladder lesions will be collected from patients who present to the study site for clinical evaluation.
  Interventions: Device: Standard High Resolution Microendoscope and/or Line-Scanning Confocal High Resolution Microendoscope

INTERVENTIONS:
Device: Standard High Resolution Microendoscope and/or Line-Scanning Confocal High Resolution Microendoscope
  Other Names: HRME and/or LSC-HRME

SUMMARY:
The goal of this study is to develop, optimize, and validate a High Resolution Imaging System in the bladder that displays images in real-time, providing automated diagnostic criteria for bladder cancer screening. High resolution images of normal bladder tissue and suspicious bladder lesions will be collected from patients who present to the study site for clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically suspicious bladder lesion or clinical finding; or who are undergoing cystoscopy as part of their routine clinical care.
* Must be willing and able to participate and provide written informed consent
* Women of childbearing age who have the possibility of being pregnant must have a negative pregnancy test prior to participation

Exclusion Criteria:

* Patient with sufficient evidence of cognitive impairment that limits the subject's ability to understand the protocol, provide informed consent, or to comply with the protocol procedures.
* Women with the possibility of having the pregnancy.
* Patients having acute infection.
* Person with Lidocaine sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified from patients who are visiting Lyndon B. Johnson Hospital (LBJ) Houston for evaluation of bladder cancer or a suspicious bladder lesion/clinical symptomatology by cystoscopy and bladder biopsy or from LBJ patients who are undergoing cystoscopy as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Specificity of Bladder Cancer Detection Imaging | baseline (at the time of imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem N Dhanani, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tang Y, Kortum A, Vohra I, Schwarz RA, Carns J, Kannady CR, Clavell-Hernandez J, Hu Z, Dhanani N, Richards-Kortum R. Initial Results of First In Vivo Imaging of Bladder Lesions Using a High-Resolution Confocal Microendoscope. J Endourol. 2021 Aug;35(8):1190-1197. doi: 10.1089/end.2020.0757. Epub 2021 Jan 21. PMID 33307957